CLINICAL TRIAL: NCT02347124
Title: Promoting Oral Health Among Tobacco Quitline Callers
Brief Title: Promoting Oral Health Among Smokers Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Consumer Wellness Solutions (Industry); University of California (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-047-E; U01DE024462-01 (NIH)
Record Dates: First submitted 2015-01-12; First posted 2015-01-27 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Oral Disease; Smoking
Keywords: smoking cessation; oral health care; tobacco quitlines
MeSH Terms: conditions — Mouth Diseases; Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care Control (Active Comparator): Standard tobacco quitline counseling program and materials + attention-matched text messaging.
  Interventions: Behavioral: Usual Care Control
- Enhanced Intervention (Experimental): Standard tobacco quitline counseling program and materials + multi-modal oral health promotion program .
  Interventions: Behavioral: Enhanced Intervention

INTERVENTIONS:
Behavioral: Usual Care Control — Standard quitline counseling and other treatment materials provided through each participating state quitline program + a series of text messages with general health promotion tips.
  Arms: Usual Care Control
Behavioral: Enhanced Intervention — Standard quitline counseling and other materials provided through each participating state quitline program + oral health-focused counseling + oral health focused text messages + access to additional oral health educational content (website and written materials) + oral health tools (toothbrush, dental floss)
  Arms: Enhanced Intervention

SUMMARY:
The current study will test the effectiveness of a multi-modal behavioral intervention (the Oral Health 4 Life program) targeted to smokers who are ready to quit smoking and seeking services through tobacco quitlines.

The investigators hypothesize that, compared to people in the control arm, participants in the enhanced intervention will:

1. Be more likely to quit smoking as evidenced by 7 day point prevalent abstinence rates at 6 month follow-up [primary outcome] and at 2 month follow-up [secondary outcome].
2. Be more likely to see a dental care professional in the past 6 months at 6 month follow-up [primary outcome].
3. Exhibit more positive change in relevant oral health knowledge/beliefs and attitudes (e.g., self-efficacy, motivation) that could influence future behavior change.

DETAILED DESCRIPTION:
Smokers (n = 722; 10 pilot participants and 712 main trial participants) will be recruited when they call to enroll in services with their state-supported tobacco quitline program. Eligible smokers who provide consent and complete the baseline assessment will be randomized to either usual care quitline intervention plus attention-matched text messaging or an enhanced program which integrates standard tobacco cessation counseling with a multi-modal, behavioral oral health promotion program.

Follow-up assessments will be conducted by phone at 2 and 6 months post-enrollment. In addition to examining primary and secondary outcomes of interest (focused on tobacco cessation and utilization of professional dental care), change in potentially relevant intermediate process measures and the incremental cost of delivering the Oral Health 4 Life program will be examined.

ELIGIBILITY:
Inclusion criteria:

* Male or female, aged 18 or older
* Eligible for multi-call services through a participating tobacco quitline managed by Alere Wellbeing
* Can read and speak in English
* Current daily smoker and smokes at least 5 cigarettes a day
* Interested in quitting smoking in next 30 days
* Have some or all natural teeth
* Have not visited a dentist for a checkup or teeth cleaning in the past 6 months and do not have an appointment scheduled in the next 6 months
* Has a cell phone capable of receiving text messages and provides cell phone number
* Has internet access for personal use
* Willing to talk about ways to improve their oral health
* Provides verbal consent to participate

Exclusion criteria:

* Self-report a diagnosis of bipolar disorder, mania, schizophrenia, dementia (e.g., has significant cognitive impairment)
* Have lived at the current address less than 6 months or plans to move in the next 6 months
* Are currently enrolled in an in-patient substance abuse treatment facility or are incarcerated
* Has a household member already enrolled in the study, based on self-report and/or mailing address on file

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McClure, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual level data.

REFERENCES:
- [Background] McClure JB, Blasi PR, Cook A, Bush T, Fishman P, Nelson J, Anderson ML, Catz SL. Corrigendum to "Oral health 4 life: Design and methods of a semi-pragmatic randomized trial to promote oral health care and smoking abstinence among tobacco quitline callers" [Contemp. Clin. Trials 57 (2017) 90-97]. Contemp Clin Trials. 2017 Oct;61:133. doi: 10.1016/j.cct.2017.07.011. Epub 2017 Jul 24. No abstract available. PMID 28750939
- [Background] McClure JB, Blasi PR, Cook A, Bush T, Fishman P, Nelson J, Anderson ML, Catz SL. Oral health 4 life: Design and methods of a semi-pragmatic randomized trial to promote oral health care and smoking abstinence among tobacco quitline callers. Contemp Clin Trials. 2017 Jun;57:90-97. doi: 10.1016/j.cct.2017.04.003. Epub 2017 Apr 12. PMID 28412230
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440
- [Derived] Blasi PR, Krakauer C, Anderson ML, Nelson J, Bush T, Catz SL, McClure JB. Factors associated with future dental care utilization among low-income smokers overdue for dental visits. BMC Oral Health. 2018 Nov 1;18(1):183. doi: 10.1186/s12903-018-0646-8. PMID 30382910

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited following registration with the Oregon (OR), Nebraska (NE), or Louisiana (LA) state quitlines. Participants were enrolled between June 2015 and July 2016.
Period: Overall Study
Arm/Group | Usual Care Control | Enhanced Intervention
Started | 360 | 358
2 Month Follow-up | 298 | 275
Completed | 267 | 259
Not Completed | 93 | 99

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Control | Enhanced Intervention | Total
Number analyzed (Participants) | 360 | 358 | 718
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (12.2) | 44.1 (12.2) | 44.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 220 | 443
  Male | 137 | 138 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 16 | 21
  Not Hispanic or Latino | 355 | 342 | 697
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Subjects were asked: "Which of the following categories best describe your race?" (may indicate all that apply).
  Categories offered were: White, Black or African-American, Native Hawaiian or Other Pacific Islander, American Indian, Other, Don't Know, Refused
  Participants
    White | 208 | 209 | 417
    Black | 113 | 95 | 208
    Other or multi-racial | 37 | 52 | 89
    Don't Know or Refused | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 360 | 358 | 718
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes] | 18.9 (9.5) | 19.3 (9.7) | 19.1 (9.7)
Last dental visit > 1 year ago [Count of Participants; unit: Participants] | 294 | 282 | 576

OUTCOME MEASURES:

1. Primary Outcome: 7 Day Point Prevalent Abstinence (PPA)
Description: 7 day point prevalent abstinence (PPA): self- report of no smoking in the past 7 days. Missing values imputed as smokers.
Time Frame: 6 month post-enrollment
Population: All participants with missing data imputed as smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 360 | 358
Participants | 109 | 121
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.13, Regression, Logistic — Adjusted for baseline sex, age, cigarettes per day, depression history, motivation, self-efficacy, current use of a stop-smoking medication, state quitline, and dental insurance; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.93 to 1.78]

2. Primary Outcome: Professional Dental Care Utilization in Past 6 Months
Description: self-reported utilization of professional dental care during study observation period
Time Frame: 6 months post-enrollment
Population: All participants with missing data imputed as not having seen a dentist.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 360 | 358
Participants | 67 | 65
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.90, Regression, Logistic — Adjusted for baseline sex, age, depression history, motivation, self-efficacy, state quitline, and dental insurance; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.69 to 1.53]

3. Secondary Outcome: 7 Day Point Prevalent Abstinence (PPA)
Description: 7 day point prevalence abstinence (PPA): self-report of no smoking in the past 7 days with missing outcomes imputed as smokers
Time Frame: 2 months post-enrollment
Population: All participants with missing data imputed as smokers.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 360 | 358
Participants | 116 | 127
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.21, Regression, Logistic — Model is adjusted for sex, age, cigarettes per day at baseline, depression, self-efficacy, motivation, self-reported use of a stop smoking medication at baseline, and stratification variables state quit line and dental insurance; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.89 to 1.69]

4. Secondary Outcome: 7 Day Point Prevalent Smoking Abstinence (PPA)
Description: Self-reported 7 day point prevalence abstinence (PPA) in complete case analysis, using respondent data only. No outcomes imputed.
Time Frame: 2 months post-enrollment
Population: Analysis limited to survey respondents (i.e., complete cases only).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 297 | 274
Participants | 116 | 127
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.04, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.01 to 2.00]

5. Secondary Outcome: 7 Day Point Prevalent Smoking Abstinence (PPA)
Description: Self-reported 7 day point prevalence abstinence (PPA) in complete case analysis. No outcomes imputed.
Time Frame: 6 months post-enrollment
Population: Complete case analysis limited to survey respondents.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 267 | 258
Participants | 109 | 121
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.09, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.95 to 1.96]

6. Other Pre Specified Outcome: Change in Oral Health Knowledge Scale Score From Baseline to 2 Month Follow up
Description: Oral health knowledge was assessed via the Brennan et al. 2010 scale, adapted from the Health Promotion and Disease Prevention Questionnaire (1985 NHIS; Corbin et al). Seven questions make up the scale:
  Seeing a dentist regularly Drinking water with fluoride Regular brushing of teeth Regular flossing of teeth Using fluoride toothpaste Avoiding sweets between meals.
  Responses and scoring to the adapted NHIS scale:
  Definitely not important = 1 Probably not important = 2 Neutral = 3 Probably important = 4 Definitely important = 5
  Scale scores are calculated by summing the responses to the 7 items, with higher scores indicating higher oral health knowledge.
  The scores have a range of 7 (minimum) to 35 (maximum).
  The study outcome is the change in this score between BL and 2 mos. The outcome is the difference in scores. A positive score indicates an increase in oral health knowledge (larger=better). A negative score indicates a decrease in knowledge.
Time Frame: Baseline to 2 months
Population: Participants providing data for this measure at the baseline and 2 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 297 | 274
scores on a scale | 0.08 (3.3) | 0.14 (3.7)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.85, Regression, Linear; Adjusted for sex, age, state quit line, and baseline knowledge score; Odds Ratio (OR) = -0.05, 95% CI 2-sided [-0.57 to 0.47]

7. Other Pre Specified Outcome: Change in Oral Health Knowledge Scale Score From Baseline to 6 Month Follow-up
Description: Oral health knowledge was assessed via the Brennan et al. 2010 scale, adapted from the Health Promotion and Disease Prevention Questionnaire (1985 NHIS; Corbin et al). Seven questions make up the scale:
  Seeing a dentist regularly Drinking water with fluoride Regular brushing of teeth Regular flossing of teeth Using fluoride toothpaste Avoiding sweets between meals.
  Responses and scoring to the adapted NHIS scale:
  Definitely not important = 1 Probably not important = 2 Neutral = 3 Probably important = 4 Definitely important = 5
  Scale scores are calculated by summing the responses to the 7 items, with higher scores indicating higher oral health knowledge.
  The scores have a range of 7 (minimum) to 35 (maximum).
  The study outcome is the change in this score between BL and 6 mos. The outcome is the difference in scores. A positive score indicates an increase in oral health knowledge (larger=better). A negative score indicates a decrease in knowledge.
Time Frame: Baseline to 6 months
Population: Participants providing data for this measure at baseline and 6 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 265 | 258
scores on a scale | -0.17 (4.0) | 0.30 (3.8)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.14, Regression, Linear; Adjusted for sex, age, state quit line, and baseline knowledge score; Odds Ratio (OR) = 0.41, 95% CI 2-sided [-0.14 to 0.96]

8. Other Pre Specified Outcome: Change in Self-efficacy (SE) for Seeing a Dentist, From Baseline to 2 Month Follow up
Description: SE to see a dentist was assessed using the following question:
  "As of today, how confident are you that you can…See a dentist in the next 6 months?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all confident", to 5="Very confident". Higher scores represented higher SE.
  The study outcome is the change in this score, between baseline and the 2-month follow-up. Therefore, the outcome is defined as the difference in score. The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in self-efficacy, and negative scores indicating a decrease in self-efficacy.
Time Frame: Baseline to 2 months
Population: Participants who provided responses to this item at baseline and 2 follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 297 | 271
scores on a scale | -0.36 (1.5) | 0.01 (1.6)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = .002, Regression, Linear; Adjusted for sex, age, state quit line, and baseline self-efficacy score; Odds Ratio (OR) = 0.35, 95% CI 2-sided [0.13 to 0.56]

9. Other Pre Specified Outcome: Change in Self-efficacy (SE) for Seeing a Dentist, From Baseline to 6 Month Follow-up
Description: SE to see a dentist was assessed using the following question:
  "As of today, how confident are you that you can…See a dentist in the next 6 months?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all confident", to 5="Very confident". Higher scores represented higher SE.
  The study outcome is the change in this score, between baseline and the 6-month follow-up. Therefore, the outcome is defined as the difference in score. The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in self-efficacy, and negative scores indicating a decrease in self-efficacy.
Time Frame: Baseline to 6 months
Population: Participants who provided responses to this item at baseline and 6 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 263 | 255
scores on a scale | -0.19 (1.5) | -0.11 (1.6)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.97, Regression, Linear — Adjusted for sex, age, state quit line, and baseline self-efficacy score; Odds Ratio (OR) = 0.00, 95% CI 2-sided [-0.22 to 0.23]

10. Other Pre Specified Outcome: Change in Motivation to Stop Smoking, From Baseline to 2 Month Follow-up
Description: Motivation to stop smoking was assessed using the following question:
  "As of today, how motivated are you to…Stop smoking for good or remain quit?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all motivated", to 5="Very motivated". Higher scores represented higher motivation.
  The study outcome is the change in this score, between baseline and the 2-month follow-up. Therefore, the outcome is defined as the difference in score.
  The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in motivation, and negative scores indicating a decrease in motivation.
Time Frame: Baseline to 2 months
Population: Participants providing responses to this item at baseline and 2 month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 297 | 273
scores on a scale | -0.17 (0.8) | -0.19 (0.9)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.16, Regression, Linear; Adjusted for sex, age, state quit line, use of stop-smoking medications, baseline motivation, and baseline cigarettes per day; Odds Ratio (OR) = -0.10, 95% CI 2-sided [-0.24 to 0.04]

11. Other Pre Specified Outcome: Change in Motivation to Stop Smoking, From Baseline to 6 Month Follow-up
Description: Motivation to stop smoking was assessed using the following question:
  "As of today, how motivated are you to…Stop smoking for good or remain quit?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all motivated", to 5="Very motivated". Higher scores represented higher motivation.
  The study outcome is the change in this score, between baseline and the 6-month follow-up. Therefore, the outcome is defined as the difference in score.
  The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in motivation, and negative scores indicating a decrease in motivation.
Time Frame: Baseline to 6 months
Population: Participants providing responses to this item at baseline and 6-month follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 263 | 256
scores on a scale | -0.37 (1.0) | -0.40 (1.0)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.83, Regression, Linear; Adjusted for sex, age, state quit line, use of a smoking cessation medication at baseline, baseline motivation score, and baseline cigarettes per day; Odds Ratio (OR) = -0.02, 95% CI 2-sided [-0.16 to 0.13]

12. Other Pre Specified Outcome: Change in Motivation for Seeing a Dentist, From Baseline to 2-month Follow-up
Description: Motivation to see a dentist was assessed using the following question:
  "As of today, how motivated are you to…see a dentist in the next 6 months?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all motivated", to 5="Very motivated". Higher scores represented higher motivation.
  The study outcome is the change in this score, between baseline and the 2-month follow-up. Therefore, the outcome is defined as the difference in score.
  The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in motivation, and negative scores indicating a decrease in motivation.
Time Frame: Baseline to 2 months
Population: Participants who provided responses to this item at baseline and 2 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 295 | 271
scores on a scale | -0.41 (1.3) | -0.19 (1.2)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.02, Regression, Linear; adjusted for sex, age, state quit line, and baseline motivation score; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.04 to 0.41]

13. Other Pre Specified Outcome: Change in Motivation for Seeing a Dentist, From Baseline to 6-month Follow-up
Description: Motivation to see a dentist was assessed using the following question:
  "As of today, how motivated are you to…see a dentist in the next 6 months?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all motivated", to 5="Very motivated". Higher scores represented higher motivation.
  The study outcome is the change in this score, between baseline and the 6-month follow-up. Therefore, the outcome is defined as the difference in score.
  The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in motivation, and negative scores indicating a decrease in motivation.
Time Frame: Baseline to 6 months
Population: Participants who provided responses to this item at baseline and 6 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 262 | 254
scores on a scale | -0.35 (1.2) | -0.27 (1.1)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.82, Regression, Linear; Odds Ratio (OR) = 0.02, 95% CI 2-sided [-0.17 to 0.21]

14. Other Pre Specified Outcome: Change in Self-efficacy (SE) for Quitting Smoking, From Baseline to 2-month Follow-up
Description: SE to quit smoking was assessed using the following question:
  "As of today, how confident are you that you can…stop smoking for good or remain quit?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all confident", to 5="Very confident". Higher scores represented higher SE.
  The study outcome is the change in this score, between baseline and the 2-month follow-up. Therefore, the outcome is defined as the difference in score.
  The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in self-efficacy, and negative scores indicating a decrease in self-efficacy.
Time Frame: Baseline to 2 months
Population: Participants who provided responses to this item at baseline and 2 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 296 | 272
scores on a scale | -0.13 (1.1) | -0.13 (1.2)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.80, Regression, Linear; Adjusted for sex, age, state quit line, baseline self-efficacy score, baseline cigarettes per day, and baseline use of stop smoking medications; Odds Ratio (OR) = -0.02, 95% CI 2-sided [-0.20 to 0.16]

15. Other Pre Specified Outcome: Change in Self-efficacy (SE) for Quitting Smoking, From Baseline to 6-month Follow-up
Description: SE to quit smoking was assessed using the following question:
  "As of today, how confident are you that you can…stop smoking for good or remain quit?"
  Responses were measured on a 5-point Likert scale ranging from 1="Not at all confident", to 5="Very confident". Higher scores represented higher SE.
  The study outcome is the change in this score, between baseline and the 6-month follow-up. Therefore, the outcome is defined as the difference in score.
  The theoretical range for the change score is -4 (minimum) to 4 (maximum), with positive scores indicating an increase in self-efficacy, and negative scores indicating a decrease in self-efficacy.
Time Frame: Baseline to 6 months
Population: Participants who provided responses to this item at baseline and 6 month follow-up.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Usual Care Control | Enhanced Intervention
Number analyzed (Participants) | 264 | 256
scores on a scale | -0.41 (1.4) | -0.34 (1.4)
Statistical Analysis 1: Comparison: Usual Care Control vs Enhanced Intervention; Test type: Superiority; p = 0.45, Regression, Linear; Adjusted for sex, age, state quit line, baseline self-efficacy score, baseline cigarettes per day, and baseline use of stop smoking medication; Odds Ratio (OR) = 0.07, 95% CI 2-sided [-0.11 to 0.26]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during each participant's active enrollment period (6 months post-randomization).
Arm/Group | Usual Care Control | Enhanced Intervention
All-Cause Mortality (participants affected / at risk) | 2/360 | 0/358
Serious Adverse Events (participants affected / at risk) | 0/360 | 3/358
Other Adverse Events (participants affected / at risk) | 11/360 | 7/358
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Control (N=360) | Enhanced Intervention (N=358)
change in heartbeat leading to ER visit. Disccontinued use of nicotien patch and resolved. (General disorders) | 0 (0) | 1 (358)
allergic reaction (General disorders) | 0 (0) | 1 (358) — Swelling of lips and tongue in response to nicotine replacement gum. Discontinued gum and symptoms resolved.
Unreversible blindness in right eye (Eye disorders) | 0 (0) | 1 (358)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care Control (N=360) | Enhanced Intervention (N=358)
Chest pain or mild tightness (General disorders) | 1 (1) | 0 (0)
Anxiety or stress, mild to moderate (General disorders) | 4 (4) | 1 (1)
Insomnia (General disorders) | 4 (4) | 1 (1)
Seizure (pre-existing disorder) (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness, mild to moderate (General disorders) | 1 (1) | 2 (2)
Behavior or mood change (while taking Zyban) (General disorders) | 0 (0) | 2 (2)
Migraine, low BP, chills and nausea (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study relied on self-reported smoking and dental care. The focus on socio-economically disadvantaged smokers limits our ability to draw conclusions about the effectiveness of the intervention if offered to higher SES smokers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/24/NCT02347124/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02347124/Prot_SAP_002.pdf